CLINICAL TRIAL: NCT04334382
Title: Hydroxychloroquine vs. Azithromycin for Outpatients in Utah With COVID-19 (HyAzOUT): A Prospective Pragmatic Trial
Brief Title: Hydroxychloroquine vs. Azithromycin for Outpatients in Utah With COVID-19
Acronym: HyAzOUT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other); Utah Department of Health (Other)
Responsible Party: Principal Investigator, Brandon Webb, Director, Transplant Infectious Diseases, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1051360
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: SARS-Co-V-2; Hydroxychloroquine; Azithromycin
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Azithromycin (Active Comparator)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine — Patients in the hydroxychloroquine arm will receive hydroxychloroquine 400mg po BID x 1 day, then 200mg po BID x 4 days (dose reductions for weight < 45kg). The drug dose (2.4 gm over 5 days) chosen falls at the lower end of doses proposed in various international trials, but it has proven in vitro efficacy, with a ratio of lung tissue trough concentrations to the EC50 (effective concentration to suppress 50% of viral activity) of >20.
  Arms: Hydroxychloroquine
Drug: Azithromycin — Patients in the azithromycin arm will receive azithromycin 500mg PO on day 1 plus 250mg PO daily on days 2-5.
  Arms: Azithromycin

SUMMARY:
This study will compare two drugs (hydroxychloroquine and azithromycin) to see if hydroxychloroquine is better than azithromycin in treating outpatients with suspected or confirmed COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Age>44 years, competent to provide consent
* Confirmed COVID-19, via a positive nucleic acid assay for COVID-19 within the last 7 days

Exclusion Criteria:

* Participants already prescribed chloroquine, hydroxychloroquine, or azithromycin
* Allergy to hydroxychloroquine or azithromycin
* History of bone marrow transplant
* Known G6PD (Glucose-6-Phosphate Dehydrogenase Deficiency) deficiency
* Chronic hemodialysis, peritoneal dialysis, continuous renal replacement therapy or Glomerular Filtration Rate < 20ml/min/1.73m2
* Liver disease (e.g. Child Pugh score ≥ B or AST (Aspartate Transaminase)>2 times upper limit)
* Psoriasis
* Porphyria
* Known cardiac conduction delay (QTc > 500mSec) or taking any prescription medications known to prolong QT interval
* Concomitant use of digitalis, flecainide, amiodarone, procainamide, or propafenone
* Prisoner
* Weight < 35kg
* Inability to follow-up - no cell phone or no address or not Spanish or English speaking
* Receipt of any experimental treatment for SARS-CoV-2 (off-label, compassionate use, or trial related) within the 30 days prior to the time of the screening evaluation
* No symptoms attributable to COVID-19
* Pregnant or nursing

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization within 14 days of enrollment | From enrollment to 14 days after enrollment
  Admitted to a hospital (not merely kept for emergency room observation)

SECONDARY OUTCOMES:
Duration of COVID-19-attributable symptoms | From enrollment to 14 days after enrollment
Hospital-free days at 28 days | Admission (day 1) to 28 days after admission (day 28)
  Hospital-free days at 28 days (number of days patient not in hospital); calculated as worst-rank ordinal with mortality by day 28 assigned the worst score
Ventilator-free days at 28 days | Admission (day 1) to 28 days after admission (day 28)
  Ventilator-free days at 28 days (number of days patient not on a ventilator); calculated as worst-rank ordinal with mortality by day 28 assigned the worst score
ICU-free days at 28 days | Admission (day 1) to 28 days after admission (day 28)
  ICU-free days at 28 days, calculated as worst-rank ordinal with mortality by day 28 assigned the worst score

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Webb, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
In order to protect patient privacy and comply with relevant regulations, identified data are unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.